CLINICAL TRIAL: NCT00179660
Title: A Phase II, Multicenter, Single-Arm, Open-Label Study To Evaluate The Safety And Efficacy Of Single-Agent Lenalidomide (Revlimid®, CC-5013) In Subjects With Relapsed Or Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: Safety And Efficacy Of Lenalidomide In Patients With Relapsed Or Refractory Aggressive Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: Prologue Research International (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-NHL-002
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Non-Hodgkins Lymphoma
Keywords: celgene; cc-5013; CC5013; NHL; Non-Hodgkins Lymphoma; Revlimid
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Lenalidomide

ARMS (1):
- Lenalidomide (Experimental): Participants received single-agent lenalidomide 25 mg orally once daily on Days 1 to 21 of every 28-day cycle for up to 52 weeks or until disease progression developed, lenalidomide treatment was discontinued for any reason, or the study was terminated.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Capsules for oral administration.
  Other Names: CC-5013; Revlimid®

SUMMARY:
To determine the activity of lenalidomide in relapsed or refractory aggressive NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age greater than or equal to 18 years at the time of signing the informed consent form
3. Able to adhere to the study visit schedule and other protocol requirements
4. Biopsy-proven non-Hodgkin's lymphoma
5. Aggressive lymphoma, the following histologies are acceptable: Follicular center lymphoma, grade 3, Diffuse large cell, Mantle cell, Transformed
6. Relapsed or refractory to previous therapy for lymphoma. Patients must have received at least one prior treatment regimen such as radiation, immunotherapy, chemotherapy, or radioimmunotherapy, and be ineligible or unwilling to undergo an autologous stem cell transplant. There is no limit on the number of prior therapies.
7. Patients must have measurable disease on cross sectional imaging that is at least 2 cm in the longest diameter.
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.
9. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug.

Exclusion Criteria:

1. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) <1,500 cells/mm^3 (1.5 x 10^9/L)
   2. Platelet count <100,000/mm^3 (100 x 10^9/L)
   3. Serum creatinine >2.5 mg/dL (221 mmol/L)
   4. Serum aspartate transaminase (AST) or alanine transaminase (ALT) >5.0 x upper limit of normal (ULN)
   5. Serum total bilirubin >2.0 mg/dL (34 mmol/L)
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
3. All patients with central nervous system (CNS) disease with the exception of those patients whose CNS disease has been treated with chemotherapy, radiotherapy or surgery and remains asymptomatic, with no active CNS disease, as shown by lumbar puncture, computed tomography (CT) scan or magnetic resonance imaging (MRI), for at least 6 months.
4. Prior history of malignancies other than non-Hodgkin's lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for > or equal to 1 year
5. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
6. Known positive for human immunodeficiency virus (HIV)
7. Pregnant or lactating females
8. Prior > or equal to grade 3 National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) allergic reaction/hypersensitivity to thalidomide
9. Prior > or equal to grade 3 NCI CTCAE rash or any desquamating (blistering) rash while taking thalidomide
10. Prior use of lenalidomide
11. Use of any standard or experimental anti-cancer drug therapy within 28 days of day 1 of study drug therapy
12. Known active Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Pacific Coast Hematology/Oncology Medical Group, Onc., Fountain Valley, California
  - UC David Cancer Center, Sacramento, California
  - Sylvester Cancer CenterUniversity Of Miami, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - New York Medical Center, MBCCOP, The Bronx, New York
  - Gunderson Clinic, Ltd, La Crosse, Wisconsin

REFERENCES:
- [Result] Wiernik PH, Lossos IS, Tuscano JM, Justice G, Vose JM, Cole CE, Lam W, McBride K, Wride K, Pietronigro D, Takeshita K, Ervin-Haynes A, Zeldis JB, Habermann TM. Lenalidomide monotherapy in relapsed or refractory aggressive non-Hodgkin's lymphoma. J Clin Oncol. 2008 Oct 20;26(30):4952-7. doi: 10.1200/JCO.2007.15.3429. Epub 2008 Jul 7. PMID 18606983

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide
Started | 50
Received Study Drug | 49
Completed 12 Cycles of Treatment | 12
Completed | 0 (Completed refers to participants ongoing in the study at the time of analysis.)
Not Completed | 50
Not completed — Adverse Event | 7
Not completed — Lack of therapeutic effect | 28
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Death | 3
Not completed — Other - Unspecified | 9

BASELINE CHARACTERISTICS:
Population: Intent to treat population includes all participants who received at least 1 dose of study drug.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White | 36
  Black | 2
  Hispanic | 10
  Asian/Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 49
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — 0 = fully active, no restrictions; 1 = restricted but ambulatory and capable of light work; 2 = ambulatory and capable of self care but unable to work.
  participants
    0 | 20
    1 | 23
    2 | 5
    Missing | 1
Non-Hodgkin's Lymphoma (NHL) Stage [Number; unit: participants] — I: The lymphoma is in only 1 lymph node area or 1 area of a single organ outside the lymph system.
  II: The lymphoma is in 2 or more groups of lymph nodes on the same side of the diaphragm, or extends from a single group of node(s) into a nearby organ.
  III: The lymphoma is found in lymph node areas on both sides of the diaphragm, or may also have spread into an area or organ next to the lymph nodes, the spleen, or both.
  IV: The lymphoma has spread outside the lymph system into an organ that is not next to an involved node or has spread to bone marrow, liver, brain, spinal cord or the pleura.
  participants
    Stage I | 1
    Stage II | 7
    Stage III | 9
    Stage IV | 32
NHL histology [Number; unit: participants]
  Follicular lymphoma grade 3 | 5
  Diffuse large B-cell lymphoma | 26
  Mantle cell lymphoma | 15
  Transformed | 3
NHL Duration [Mean (Standard Deviation); unit: years] | 4.0 (4.91)
International Prognostic Index (IPI) [Number; unit: participants] — A clinical tool to aid in predicting the prognosis of patients with aggressive NHL. One point is assigned for each of the following risk factors:
  * Age greater than 60 years
  * Stage III or IV disease
  * Elevated serum lactate dehydrogenase
  * ECOG performance status of 2, 3, or 4 -> 1 extranodal site
  The sum of the points allotted correlates with the following risk groups:
  Low risk (0-1 points): 5-year survival of 73% Low-intermediate risk (2 points): 5-year survival of 51% High-intermediate risk (3 points): 5-year survival of 43% High risk (4-5 points): 5-year survival of 26%
  participants
    Low (0 to 1) | 8
    Low/Intermediate (2) | 22
    High/Intermediate (3) | 13
    High (4 to 5) | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response
Description: Response was defined as participants with a complete response (CR), unconfirmed complete response (Cru) or partial response (PR), assessed using the International Workshop Lymphoma Response Criteria (IWLRC) and based on best responses as determined by the investigator.
  CR: Complete disappearance of all detectable clinical and radiographic evidence of disease, disappearance of any disease-related symptoms, and normalization of biochemical abnormalities.
  Cru: Criteria for CR above but with 1 or more of the following:
  * A residual lymph node mass > 1.5 cm in greatest transverse diameter that has regressed by more than 75% in the sum of the products of diameters (SPD)
  * Indeterminate bone marrow (increased number or size of aggregates without cytologic or architectural atypia).
  PR: 50% decrease in SPD of the 6 largest dominant nodes or nodal masses. No increase in the size of other nodes, liver, or spleen. Splenic and hepatic nodules must regress by at least 50% in the SPD.
Time Frame: From enrollment through study completion. Median duration on study was 3.7 months, with a maximum of 32.5 months.
Population: Intent-to-treat (ITT) population, which included all enrolled patients who received at least 1 dose of study drug. Patients who dropped out without having a response assessment or who had a response after they had received other anti-cancer treatments were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 49
percentage of participants | 34.7 [21.7 to 49.6]

2. Secondary Outcome: Percentage of Participants With Tumor Control
Description: Tumor control was defined as participants with a complete response, unconfirmed complete response, partial response or stable disease (SD), assessed using the International Workshop Lymphoma Response Criteria (IWLRC) and based on best responses as determined by the investigator.
  SD was defined as a response less than a PR (see above) but not Progressive Disease (PD).
  PD was defined as
  * ≥ 50 % increase from nadir in the SPD of any previously identified abnormal node for partial responders or non-responders.
  * Appearance of any new lesion during or at the end of therapy.
Time Frame: From enrollment through study completion. Median duration on study was 3.7 months, with a maximum of 32.5 months.
Population: Intent-to-treat (ITT) population. Patients who dropped out without having a response assessment or who had a response after they had received other anti-cancer treatments were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 49
percentage of participants | 59.2 [44.2 to 73.0]

3. Secondary Outcome: Duration of Response
Description: The duration of response was calculated as the first response assessment demonstrating evidence of at least a partial response to the first documentation of progressive disease (as determined by computed tomography scan) or death due to NHL, whichever occurred first. For participants without documentation of progression, the duration of response was censored at the last date of tumor assessment indicating no progression. Median was based on the Kaplan-Meier estimate.
Time Frame: From enrollment through study completion. Median duration on study was 3.7 months, with a maximum of 32.5 months.
Population: Intent to treat population with a response = CR, CRu or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 17
months | 10.2 [4.0 to 16.3]

4. Secondary Outcome: Duration of Tumor Control
Description: The duration of tumor control was calculated as the time from the first response assessment demonstrating at least stable disease to the first documentation of progressive disease or death due to NHL. For participants without documentation of progression, the duration of response was censored at the last date of tumor assessment indicating no progression. Median was based on the Kaplan-Meier estimate.
Time Frame: From enrollment through study completion. Median duration on study was 3.7 months, with a maximum of 32.5 months.
Population: Intent to treat population with tumor control (CR, CRu, PR or SD).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 29
months | 6.0 [2.9 to 11.1]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the start of study drug therapy to the first observation of disease progression or death due to any cause, whichever came first.
  Participants who withdrew for any reason or received another NHL therapy including stem cell transplantation without documented progressive disease were censored on the date of their last adequate response assessment indicating no progression (or last adequate assessment prior to receiving other NHL therapy). Participants who were still active without progressive disease at the time of the data cut-off date were censored on the date of their last adequate response assessment.
Time Frame: From enrollment through study completion. Median duration on study was 3.7 months, with a maximum of 32.5 months.
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 49
months | 3.6 [2.0 to 6.3]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The Investigator determined the relationship between the administration of study drug and the occurrence of an AE as suspected if the temporal relationship of the adverse event to study drug administration made a causal relationship possible, and other drugs, therapeutic interventions, or underlying conditions did not provide a sufficient explanation for the observed event.
  The Investigator graded the severity of AEs according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria and the following scale:
  * Grade 1 = Mild
  * Grade 2 = Moderate
  * Grade 3 = Severe
  * Grade 4 = Life threatening
  * Grade 5 = Death
  A Serious AE is defined as any AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or constitutes an important medical event.
Time Frame: From the start of study drug through 30 days after the last dose of study drug. Maximum time on study drug was 15.2 months.
Population: Safety Population, which includes all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 49
participants
  Any adverse event | 49
  Adverse event related to study drug | 42
  Grade 3-5 adverse event | 36
  Grade 3-5 adverse event related to study drug | 27
  Serious adverse event | 21
  Serious adverse event related to study drug | 6
  AE leading to discontinuation of study drug | 9
  Related AE leading to study drug discontinuation | 4
  AE leading to dose reduction or interruption | 28

ADVERSE EVENTS:
Time Frame: From the start of study drug through 30 days after the last dose of study drug. Maximum time on study drug was 15.2 months
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 21/49
Other Adverse Events (participants affected / at risk) | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=49)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Anemia NOS (Blood and lymphatic system disorders) | 1
Coombs positive hemolytic anemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Abdominal pain NOS (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Chest pain (General disorders) | 1
Malaise (General disorders) | 1
Autoimmune disorder NOS (Immune system disorders) | 1
Pneumonia NOS (Infections and infestations) | 3
Bronchopneumonia NOS (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Osteomyelitis NOS (Infections and infestations) | 1
Sepsis NOS (Infections and infestations) | 1
Staphylococcal bacteremia (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Non-Hodgkin's lymphoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Breast cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cauda equina syndrome (Nervous system disorders) | 1
Convulsions NOS (Nervous system disorders) | 1
Spinal hematoma (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Sweating increased (Skin and subcutaneous tissue disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=49)
Fatigue (General disorders) | 19
Pyrexia (General disorders) | 8
Oedema Peripheral (General disorders) | 6
Pain NOS (General disorders) | 3
Constipation (Gastrointestinal disorders) | 15
Diarrhoea NOS (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 10
Abdominal Pain NOS (Gastrointestinal disorders) | 4
Vomiting NOS (Gastrointestinal disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Anaemia NOS (Blood and lymphatic system disorders) | 15
Leukopenia NOS (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 8
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypermagnesaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 5
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 5
Peripheral Neuropathy NOS (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Neuropathy NOS (Nervous system disorders) | 3
Rash NOS (Skin and subcutaneous tissue disorders) | 13
Night Sweats (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3
Platelet Count Decreased (Investigations) | 11
Neutrophil Count Decreased (Investigations) | 9
White Blood Cell Count Decreased (Investigations) | 9
Haemoglobin Decreased (Investigations) | 8
Alanine Aminotransferase Increased (Investigations) | 4
Aspartate Aminotransferase Increased (Investigations) | 3
Blood Alkaline Phosphatase NOS Increased (Investigations) | 3
Blood Creatinine Increased (Investigations) | 3
Infection NOS (Infections and infestations) | 4
Upper Respiratory Tract Infection NOS (Infections and infestations) | 4
Urinary Tract Infection NOS (Infections and infestations) | 3
Insomnia (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally thirty (60) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.